CLINICAL TRIAL: NCT06623175
Title: Effects of Acupuncture in Spontaneous Rapture of Membranes: Applicability and Effectiveness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Fabio Facchinetti (Other)
Responsible Party: Sponsor-Investigator, Prof. Fabio Facchinetti, Professor, University of Modena and Reggio Emilia
Organization: University of Modena and Reggio Emilia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 126/2018
Record Dates: First submitted 2024-09-24; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: PROM (Pregnancy); Induced; Birth; Acupuncture; Labour; Cervical Ripening
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Acupuncture group (Experimental): This group of patients were randomly assigned to receive acupuncture in the first 24h after PROM, consisting in the insertion of sterile disposable acupuncture needles, stimulating specific acupoints able to enhance uterine activity, ripe the cervix and reduce anxiety.
  Interventions: Device: Acupuncture needles
- Non acupuncture group (No Intervention): This group of patients were randomly assigned to the no acupuncture group, meaning they received no intervention in the first 24h after PROM.

INTERVENTIONS:
Device: Acupuncture needles — See arm description
  Arms: Acupuncture group

SUMMARY:
The aim of the study is to investigate the effects of acupuncture in women presenting with spontaneous rapture of membranes (PROM) at term and negative swab for Streptococcus Agalactie to promote a spontaneous onset of labour and avoid labour induction after 24 hours, accordingly to our policy. Secondary outcomes were considered the duration of first and second stage of labour, the time elapsed between PROM and delivery.

ELIGIBILITY:
Inclusion Criteria:

* PROM after 37 weeks of gestation
* absence of maternal and fetal complications
* negative swab of Streptococcus Agalactiae
* limpid amniotic fluid
* absence of uterine contractions after 6 hours of observation
* single pregnancy

Exclusion Criteria:

* PROM before 37 weeks of gestation
* presence of maternal and fetal complications
* positive swab of GBS
* M1 - M3 amniotic fluid
* regular uterine contractions during the first 6 hours of observation
* twin pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Rate of spontaneous onset of labour and avoidance of labour induction after 24 hours from PROM | Time between PROM and birth/delivery

SECONDARY OUTCOMES:
Duration of second stage of labour | Time between established labour and delivery
Time elapsed between PROM and delivery | Time elapsed between PROM and delivery
Duration of first stage of labour | Time between PROM and active labour

OTHER OUTCOMES:
Time elapsed between PROM and full dilation | Time elapsed between PROM and full dilation (10 cm)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero-Universitaria di Modena, Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/8912994/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/2216201/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/2187524/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/28050900/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/28121831/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/9396886/
- See also: Related Info — https://salute.regione.emilia-romagna.it/normativa-e-documentazione/linee-di-indirizzo/archivio-documenti-tecnici/linee-guida/linee-guida-sulla-sorveglianza-del-benessere-fetale-nel-travaglio-del-parto
- See also: Related Info — https://www.saperidoc.it/flex/cm/pages/ServeBLOB.php/L/IT/IDPagina/1440
- See also: Related Info — https://www.hoepli.it/libro/atlante-di-agopuntura/9788820325176.html
- See also: Related Info — https://www.hoepli.it/libro/obstetrics-and-gynecology-in-chinese-medicine/9780443104220.html
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/69288/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/10406751/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32032444/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29036756/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/9692336/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/11802511/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/14685931/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/15673989/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/19757334/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/25911499/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/17091416/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/17963050/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4586896/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/6507532/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/1630743/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/9917943/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/8912990/